CLINICAL TRIAL: NCT04425226
Title: Safety and Efficacy Study of Pembrolizumab in Combination With LENvatinib in Participants With Hepatocellular Carcinoma (HCC) Before Liver Transplant as Neoadjuvant TherapY--PLENTY Randomized Clinical Trial
Brief Title: Pembrolizumab and LENvatinib in Participants With Hepatocellular Carcinoma (HCC) Before Liver Transplant
Acronym: PLENTY202001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Renji-IIT-2020-0005
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Liver Transplant; Complications; Hepatocellular Carcinoma Recurrent
MeSH Terms: interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab plus Lenvatinib (Experimental): Participants receive intravenous (IV) pembrolizumab at 200 mg on Day 1 of each 21-day cycle. Number of cycles: until >42 days before liver transplantation or unacceptable toxicity develops. Patients receive Lenvatinib 8-12mg(basing on weight), once a day, oral at least 38 days of each 6 weeks cycle until >7 days before liver transplantation.
  Interventions: Drug: Pembrolizumab Injection [Keytruda]; Drug: Lenvatinib Oral Product
- Comparator (No Intervention): Participants are advised to stay as healthy as possible and wait regularly

INTERVENTIONS:
Drug: Pembrolizumab Injection [Keytruda] — Pembrolizumab (Keytruda, MSD China) is a recombinant anti-human PD-1 monoclonal antibody.
  Other Names: Keytruda; MK-3475; Pembrolizumab
  Arms: Pembrolizumab plus Lenvatinib
Drug: Lenvatinib Oral Product — Lenvatinib (Lenvima, Eisai China) is a novel angiogenesis inhibitor which targets vascular endothelial growth factor 1-3, fibroblast growth factor receptor 1-4, platelet-derived growth factor receptor β, RET and KIT
  Other Names: LENVIMA; Lenvatinib
  Arms: Pembrolizumab plus Lenvatinib

SUMMARY:
Objectives of Study：This study will evaluate the safety and efficacy of pembrolizumab in combination with lenvatinib as neoadjuvant therapy in participants with hepatocellular carcinoma (HCC) exceeding Milan criteria before liver transplant.

The primary hypothesis of this study are that neoadjuvant pembrolizumab plus lenvatinib is superior to regularly waiting in the list with respect to: 1) recurrence-free survival (RFS) as assessed by blinded independent central review (BICR); and 2) Objective Response Rate (ORR).The investigators design a clinical study to explore whether the combination above as a neoadjuvant treatment in patients with advanced HCC before liver transplant could reduce postoperative recurrence and to analyze potential immune biomarker of therapeutic response.

DETAILED DESCRIPTION:
Participates would be randomly assigned (1:1) to experimental or Comparator/Control by computer-generated allocation based on the envelope method and the hierarchical block randomization method(hierarchy: BCLC stage and AFP level). The envelopes are sealed opaque, and sequentially numbered.Randomization is performed by the trial coordinator.The random number table and the block assignment number table will be kept confidential by the full-time secretary of this project.Center-stratified block-permuted randomization is used in this trial. Then permuted block randomization is used for each stratum with a block size of 4.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically or cytologically or by radiological criteria proven hepatocellular carcinoma（exceeding Milan criteria）; known mixed histology (e.g. hepatocellular carcinoma plus cholangiocarcinoma) or fibrolamellar variant is not allowed
* Has an eligibility scan (CT of the chest, triphasic CT scan or MRI of the abdomen, and CT or MRI of the pelvis) <1 week before the treatment of pembrolizumab in combination with lenvatinib. Randomization needs to occur within 1 weeks after recruitment in the waiting list.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days prior to Cycle 1, Day 1.
* Has a Child-Pugh A-B7 liver score (5 to 7 points) within 7 days prior to Cycle 1, Day 1.
* Has controlled hepatitis B (Hep B)
* The estimate time length between enrollment and liver transplantation should be at least 3 months
* No prior systemic therapy, local therapy (TACE etc.)>6w
* If female, is not pregnant or breastfeeding, and at least one of the following conditions applies: 1) Is not a woman of childbearing potential (WOCBP); or 2) Is a WOCBP and using a contraceptive method that is highly effective or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (a WOCBP must have a negative pregnancy test within 72 hours before the first dose of study treatment).
* Has adequate organ function.
* Granulocytes >= 1,500/uL
* Hemoglobin >= 8.5 g/dL; patients with recent or ongoing gastrointestinal bleed may not be transfused to reach the entry hemoglobin of 8.5 g/dL; physicians should ensure patients requiring transfusion prior to registration do not have an occult or clinically apparent gastrointestinal bleed
* Platelets >= 75,000/uL
* Creatinine =< 1.5 x upper limit of normal (ULN) (or creatinine clearance calculated >= 60 cc/minute)
* Bilirubin =< 3 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 5 x ULN
* Prothrombin time (PT)-international normalized ratio (INR) =< 1.7 (not required for patients on anticoagulation agents; patients who are being therapeutically anticoagulated with an agent such as Coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists)
* Patients with a history of hypertension should be well controlled (< 140/90 mmHg) on a regimen of anti-hypertensive therapy
* Significant history of cardiac disease is not allowed:
* Congestive heart failure > class II New York Heart Association (NYHA) Myocardial infarction within 6 months prior to registration Serious myocardial dysfunction, defined as scintigraphically (multigated acquisition scan [MUGA], myocardial scintigram) determined absolute left ventricular ejection fraction (LVEF) below 45% or an LVEF on echocardiogram (ECHO) below the normal limit at the individual institution

Exclusion Criteria:

* Surgery within the past 3 years.
* Has had esophageal or gastric variceal bleeding within the last 6 months.
* Has clinically apparent ascites on physical examination.
* Has had clinically diagnosed hepatic encephalopathy in the last 6 months.
* Has received liver ablation, radiofrequency or microwave ablation, radiotherapy in the last 6 months.
* Has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy.
* Has dual active Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) infection at study entry.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has known active tuberculosis (TB; Bacillus tuberculosis).
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Has received prior systemic anti-cancer therapy for HCC including investigational agents.
* Is receiving any of the following prohibited concomitant therapies:1) Antineoplastic systemic chemotherapy or biological therapy; 2) Immunotherapy not specified in this protocol; 3) Investigational agents other than pembrolizumab; 4) Radiation therapy; 5) Oncological surgical therapy; or systemic glucocorticoids for any purpose other than to modulate symptoms from an AE that is suspected to have an immunologic etiology.
* Has received a live vaccine within 30 days prior to the first dose of study treatment.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to Cycle 1, Day 1.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to Cycle 1, Day 1.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to ~4 years
  RFS is defined as the time from randomization to first documentation of disease recurrence (local, regional, or distant) as assessed by BICR or by pathology consistent with HCC if required per the site's standard of care, or death due to any cause (both cancer and non-cancer causes of death)

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | one year
  Proportion of patients whose tumor volume control (reduced or enlarged) reaches a predetermined value and can maintain a minimum time limit.
Percentage of Participants who Experience an Adverse Event (AE) | one year
  An AE is defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy can be determined.
Percentage of Participants who Discontinue Study Treatment due to an AE | Up to ~1 year
  An AE is defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy can be determined.
Objective Response Rate (ORR) | one year
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Xia, MD., Ph.D., Study Chair — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU; Hao Feng, MD., Ph.D., Principal Investigator — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China